CLINICAL TRIAL: NCT00907465
Title: Measurement of Sedentary Behavior in African American Adults
Brief Title: Sedentary Behavior in African Americans
Acronym: SeBA
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Robert Newton, Principal Investigator, Pennington Biomedical Research Center
Other Study IDs: PBRC 27013; 1K01HL088723-01 (NIH)
Record Dates: First submitted 2009-05-18; First posted 2009-05-22 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-12

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Calibration study: These individuals were used to develop cut points for sedentary behavior using accelerometers and a metabolic chamber.

SUMMARY:
The study is designed to develop methods for objectively measuring sedentary behavior, assess the association between objectively measured sedentary behavior and cardiovascular disease outcomes, and develop an intervention to reduce sedentary behavior, in African American adults.

ELIGIBILITY:
Inclusion Criteria:

* self-classify yourself as African American
* are aged 18 years or older
* are free of serious medical condition, such as cancer, cardiovascular disease, or emphysema.
* are free of serious medical conditions that would prevent participant from engaging in physical activity.
* are willing to have a scan completed that measures your body composition
* are willing to stay in metabolic chamber for 8.5 hours (8:00am until 4:30 pm)
* are willing to wear an accelerometer for 2, one-week periods following your chamber stay. There will be one week in-between the 2, one-week periods.
* are willing to complete questionnaire related to your level of activity
* weigh less than 250 lbs.

Exclusion Criteria:

* unwilling or unable to perform activities in protocol
* on medications
* a woman who is intending to become pregnant, or who is pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community members of Baton Rouge, LA.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2007-07; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Sedentary behavior | 2009-2010

SECONDARY OUTCOMES:
Blood pressure | 2009-2010
High density lipoproteins | 2009-2010

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Newton, Ph.D., Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States